CLINICAL TRIAL: NCT05409365
Title: Assessment of Squamous Cell Carcinoma antigen2 in Verruca Vulgaris
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fatma Aboelmaged Abdelgaber, Resident of Dermatology and Venereology, Sohag University
Other Study IDs: Soh-Med-22-04-07
Record Dates: First submitted 2022-06-01; First posted 2022-06-08 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Verruca Vulgaris; Healthy
MeSH Terms: conditions — Warts | interventions — leupin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Immunohistochemical staining monoclonal antibodies to SCCA2 (SERPINB4/ SCCA2 antibody) — Immunohistochemical staining

SUMMARY:
This study aims to assess the expression of SCCA2 in the skin of patients with warts and to detect its correlation with characteristics of warts.

DETAILED DESCRIPTION:
Type of the study: Cross sectional study. Patients: This study will include 25 patients with verruca vulgaris and 25 healthy volunteers.

Inclusion criteria:

Patients present with warts (verruca vulgaris type).

Exclusion criteria:

Subjects who presenting with allergic diseases or other dermatological diseases or had a history of squamous cell carcinoma will be excluded from this study One skin biopsy will be taken from each healthy volunteers of the control group via 2-mm disposable punches under complete sterile precautions. Two biopsies will be taken from patients with wart lesion one from verruca vulgaris via 5-mm disposable punches and another from non-affected skin via 2-mm disposable punches under complete sterile precautions.

Biopsy handling: Each specimen in both groups will be fixed in formalin and embedded in paraffin to form paraffin blocks. Serial sections will be obtained from each block and stained with hematoxylin and eosin (H&E) for histological diagnosis.

Stained sections will be examined under a light microscope. To confirm the diagnosis of wart, the grade of inflammation and the density of dermal inflammatory infiltrate will be classified as follows Grade 0, no infiltrate; Grade 1, mild; Grade 2, moderate; or Grade 3, marked infiltrate.

Immunohistochemical staining: investigators will use monoclonal antibodies to SCCA2 (SERPINB4/ SCCA2 antibody). Immunohistochemical staining will be performed the pattern of immunostaining for SCCA2 will be evaluated in both the epidermis and dermis of wart lesions. The immunohistochemical score (IHC) range will be as follows: 0: negative expression of SCCA2; 1+: weak expression of SCCA2; 2+: moderate expression of SCCA2; and 3+: strong expression of SCCA2.

ELIGIBILITY:
Inclusion Criteria:

* Patients present with warts (verruca vulgaris type).

Exclusion Criteria:

* Subjects who presenting with allergic diseases or other dermatological diseases or had a history of squamous cell carcinoma will be excluded from this study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Squamous Cell Carcinoma Antigen2 in Verruca Vulgaris | through study completion, an average of 1 year
  Immunohistochemical staining: investigators will use monoclonal antibodies to SCCA2 (SERPINB4/ SCCA2 antibody). Immunohistochemical staining will be performed the pattern of immunostaining for SCCA2 will be evaluated in both the epidermis and dermis of wart lesions. The immunohistochemical score (IHC) range will be as follows: 0: negative expression of SCCA2; 1+: weak expression of SCCA2; 2+: moderate expression of SCCA2; and 3+: strong expression of SCCA2.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Ahmed Abd El-Latif Abd El-Latif, Lecturer, Study Director — Director
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided